CLINICAL TRIAL: NCT01113359
Title: The Potential Link Between HCMV Infection and Essential Hypertension
Brief Title: The Link Between Human Cytomegalovirus (HCMV) and Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Jun Cai / Heart Center, Beijing Chao Yang Hospital
Other Study IDs: BJCY-CV-2010001; YXinchun (Registry Identifier: YXinchun)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2010-04

CONDITIONS: HCMV Infection; Hypertension
Keywords: HCMV infection; Hypertension; The Potential Link Between HCMV Infection and Essential Hypertension
MeSH Terms: conditions — Cytomegalovirus Infections; Hypertension; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: hypertensive patients
- control group: healthy volunteer

SUMMARY:
It has been reported that mouse cytomegalovirus infection alone can elevate the blood pressure in mice. Since HCMV has uniquely evolved with its human host, with little genetic similarity to the animal CMV counterparts, and it only replicates in human, an epidemiological study is required to define the relevance of HCMV infection and expression of hcmv-miRNA-UL112 to the pathogenesis of essential hypertension.

The investigators found that hcmv-miR-UL112, a human cytomegalovirus (HCMV)-encoded miRNA, was highly expressed in the hypertensive patients. Among the top miRNA target predictions, the investigators demonstrate that IRF-1 is a direct target gene of hcmv-miR-UL112, along with MICB that has been previously reported. Both IRF-1 and MICB play critical roles in immuno/inflammatory and anti-infection response. Thus, the investigators speculated that IRF-1 and MICB repression by hcmv-miR-UL112 could be considered a unifying mechanism that evades the host response at several levels: antiviral, inflammatory, and immune. In addition, there is an increasing evidence that IRF-1 may be important in apoptosis, angiogenesis, neointima formation and the pathogenesis of vascular diseases. IRF-1 can up-regulate angiotensin II type 2 receptor (AGTR2) that exerts antiproliferative and proapoptotic actions and affects regulation of blood pressure. It has been reported that the targeted disruption of the mouse AGTR2 gene resulted in a significant increase in blood pressure and increased sensitivity to angiotensin II. The nitric oxide synthase expression and NO synthesis in macrophages and distinct cardiomyocytes are induced and controlled by IRF-1 in response to inflammation, important steps in vascular biology that may improve endothelial function and inhibit smooth muscle cell migration, and a key pathophysiological event in hypertension. Collectively, these reports support a strong relationship between IRF-1 regulation and hypertension, indicating a potential role of hcmv-miR-UL112 and HCMV infection in the pathogenesis of hypertension.Thus, the investigators want to investigate the potential link between HCMV infection and essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension are assessed for potential secondary causes, for the severity of hypertension, other risk factors and for end-organ damage
* Aged between 30 to 60 years
* Untreated (whole day average > 140/90 mmHg) or treated hypertension whole-day average < 140/85), as determined by 24-hour blood pressure monitoring.

Exclusion Criteria:

* Cancer
* Diabetes
* Smoking
* Renal failure
* Stroke
* Peripheral artery disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: essential hypertensive patients:
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The positive rate of HCMV infection in hypertensive patients and healthy control | 1 month

SECONDARY OUTCOMES:
HCMV copies number per ml plasma of hypertensive patients and healthy controls | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Xin-Chun Yang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Jun Cai, Beijing, Chaoyang, China